CLINICAL TRIAL: NCT05224388
Title: Evaluating Dose Regimen of Intravenous Unfractionated Heparin and Low Molecular Weight Heparin in Critical Ill Patients Versus Critical Ill COVID-19 Patients Using Anti-Xa Levels.
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07991
Record Dates: First submitted 2022-02-03; First posted 2022-02-04 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Deep Vein Thrombosis; Anticoagulants and Bleeding Disorders; Critical Illness
MeSH Terms: conditions — COVID-19; Venous Thrombosis; Hemostatic Disorders; Critical Illness | interventions — Enoxaparin; Heparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Critically ill, prophylactic dose regimen: Prophylaxis of deep vein trombosis in critically ill patients
  Interventions: Drug: Enoxaparin; Drug: Heparin
- Critically ill, therapeutic dose regimen: Therapeutic anticoagulation for tromboembolic pathology in critically ill patients
  Interventions: Drug: Enoxaparin; Drug: Heparin
- Covid, prophylactic dose regimen: Prophylaxis of deep vein trombosis in Covid patients
  Interventions: Drug: Enoxaparin; Drug: Heparin
- Covid, therapeutic dose regimen: Therapeutic anticoagulation for tromboembolic pathology in Covid patients
  Interventions: Drug: Enoxaparin; Drug: Heparin

INTERVENTIONS:
Drug: Enoxaparin — Use of enoxaparin in either prophylactic dose regimen or therapeutic dose regimen
  Other Names: Clexane
Drug: Heparin — Use of heparin in either prophylactic dose regimen or therapeutic dose regimen

SUMMARY:
To see whether our increased dosing regimen of unfractionated heparin (UF) and low molecular weight heparin (LMWH) in COVID-19 patients was effective at preventing thrombo-embolic complications. We did regular anti-Xa tests to optimise the dose of our thromboprophylaxis. Furthermore, we want to examine the time it takes to reach adequate anti-Xa levels, to determine additional risk factors and do a subgroup analysis. Lastly, we will study if there are possible complications of our thromboprophylactic therapy.

DETAILED DESCRIPTION:
COVID-19 took the world by storm with its fast spread, high number of infected patients and its potential to range from mild illness to very severe respiratory distress. This pandemic is currently the focus of a lot of research, however there are still a lot of unknowns regarding COVID-19. Current literature shows that COVID-19 patients have an increased risk for thrombo-embolic events which is why patients at the Ghent university hospital get increased dose of thrombo-prophylactic therapy. Patients were also screened for presence of deep venous thrombosis using ultrasound.

Anti-Xa is a test in which the we determine the activity of the antithrombine-heparine complex on factor Xa. Using this test allowed us to measure the effect of our UF of LWMH and adjust the dose if needed.

At this moment It is still unclear how high the prevalence of thromboembolic events in this group of patients is and whether our thromboprophylaxic therapy prevents this. We also looked into the time it took for anti-Xa to reach adequate levels in our dosing regimen. Furthermore, current risk factors for thromboembolic complications in COVID-19 patients are still unclear. We compared the results of the COVID-19 patients to a group of critical ill patients without COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Hospitalisation required
* ICU admission

Exclusion Criteria:

* Coagulopathies prior to COVID 19 infection (known thromboembolism in the last 6 months i.e. deep venous thrombosis, pulmonary embolism, …)
* Therapeutic anticoagulation on moment of ICU admission
* Major trauma
* Major bleeding
* Cerebro vascular accident or neuro trauma in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients and other critical ill patients, during their stay in the intensive care unit of the Ghent University Hospital.
Sampling Method: Probability Sample
Enrollment: 813 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluate dose regimen of UFH en LMWH for critically ill patients and Covid-19 patients in: - preventing thrombo-embolic complications - time to reach adequate prophylactic antiXa range | 36 hours
  36 hours after start of the intervention drug (enoxaparin or heparin) the antiXa level is measured

SECONDARY OUTCOMES:
Possible risk factors for thrombo-embolic complications in COVID-19 patients | Time of discharge or death
  Risk factors are minor bleeding, major bleeding
Safety of increased dose of thromboprophylaxis in Covid-19 patients | Time of discharge or death
  Special consideration of minor or major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Harlinde Peperstraete, MD, Study Chair — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided